CLINICAL TRIAL: NCT03099538
Title: Ixekizumab in the Treatment of Bullous Pemphigoid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Aaron R. Mangold, Assistant Professor of Dermatology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#16-008302
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Bullous Pemphigoid; Pemphigoid
Keywords: Ixekizumab; Bullous Pemphigoid; Pemphigoid; IL17; IL-17; Interleukin 17
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — ixekizumab

STUDY DESIGN:
Intervention Model Description: This is a single center, exploratory, open-label, single-arm design study of 12 patients with BP. Treatment naïve and treatment refractory patients with BP will be treated with Ixekizumab. Patients who are non-responders, to physician choice standard of care, will undergo a washout period and will be enrolled in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ixekizumab (Experimental): Ixekizumab subcutaneous 160mg week 0, 80mg weeks 2, 4, 6, 8, 10, 12.
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Ixekizumab — Subcutaneous injection
  Other Names: Taltz

SUMMARY:
Recently, Interleukin (IL)-17 has been identified as a key driver of chronic inflammation in Bullous Pemphigoid (BP). Ixekizumab is a recombinant high-affinity fully human monoclonal antibody that targets IL-17A Immunoglobulin gamma-1 (IgG1)/kappa-class. The purpose of this study is to determine the effect of Ixekizumab on BP patients.

DETAILED DESCRIPTION:
BP is the most common auto-immune blistering disease of the skin and causes significant morbidity. BP disproportionally affects the elderly population and the current, non-specific immunosuppressive therapies, in addition to patient comorbidities, are associated with a high risk of infection related mortality. Neutrophils and their proteases have been shown to play a major role in the cleavage of Bullous Pemphigoid 180 Antigen (BP180) in BP. Mast cells and other cellular mediators also contribute to the pro-inflammatory environment within and surrounding blisters of BP. However, the prior targeting of mast cells and basophils has resulted in unpredictable disease control. Recently, IL-17 has been identified as a key driver of chronic inflammation in BP. With the increasing aged population in the United States, BP will increase in prevalence and the development of a more targeted approach will be necessary to decrease morbidity and mortality. IL-17 inhibition with Ixekizumab may have targeted, disease-modifying effects on BP. The primary objective is to test the effect of Ixekizumab in the treatment of the autoimmune blistering disease, BP.

ELIGIBILITY:
Subjects eligible for inclusion in this study have to fulfill all of the following Inclusion criteria:

* Subjects must be able to understand and comply with the requirements of the study and communicate with the investigator. Subjects must give written, signed, and dated informed consent before any study related activity is performed. When appropriate, a legal representative will sign the informed consent according to local laws and regulation
* Both men and women must be at least 18 years of age at the time of screening
* Subjects must have clinical, histological, and serological features of BP
* Urticarial plaques and/or vesicles and bullae
* Characteristic eosinophilic spongiosis and/or subepidermal separation of the skin
* Positive direct immunofluorescence (IgG and or C3 at the basement membrane zone) or indirect immunofluorescence (IgG on the roof of salt- split skin) or positive serologies on ELISA for BPAG1 or BPAG2
* Subjects must have treatment naive BP or treatment refractory disease, as defined by failure of at least one established treatment for BP
* Candidate for systemic therapy, defined by
* involvement of greater than 5 percent body surface area or moderate to extensive disease as defined by: the mean number of new bullae and urticarial plaques that have appeared over the course of 3 days as determined by the investigator or referring physician (moderate disease defined by greater than 1 and less than 10 new bullae and greater than 5 urticarial plaques and extensive disease by greater than 10 new bullae)
* Failure of prior therapy
* Topical treatment
* Systemic immunosuppressant
* Oral antibiotics and/or niacinamide

Exclusion Criteria:

Subjects fulfilling any of the following criteria are not eligible for inclusion in this study. In order to ensure the recruitment of a representative sample of all eligible subjects, the investigator may apply no additional exclusions.

* Forms of BP other than classic BP (e.g. mucous membrane BP, Brunsting-Perry BP, p200 BP, p105 BP, or BP with concomitant pemphigus vulgaris Drug-induced BP (e.g., new onset or current exacerbation from angiotensin converting enzyme inhibitors, penicillamine, furosemide, phenacetin)
* Subjects who are receiving treatments known to worsen BP and use of penicillamine or phenacetin and those on angiotensin converting enzyme inhibitors or furosemide who have not been on a stable dose at least 4 weeks prior to enrollment.
* Ongoing use of prohibited treatments.
* Previous exposure to Ixekizumab or any other biologic drug directly targeting IL-17A or IL-17 (receptor A)RA
* Use of any other investigational drugs within 5 half-lives of the investigational treatment before study drug initiation or until the pharmacodynamics effect has returned to baseline, whichever is longer
* Previous use of IL-20 monoclonal antibody
* Pregnant or nursing (lactating) women (pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test)
* Women of childbearing potential [Post-menopausal or not of child-bearing potential is defined by: 1 year of natural (spontaneous) amenorrhea or Surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks ago. Oophorectomy alone must confirmed by follow up hormone level assessment to be considered not of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception which includes:
* Total abstinence (Periodic abstinence and withdrawal are not acceptable methods of contraception)
* Female sterilization (bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment. Oophorectomy alone requires follow up hormone level assessment for fertility.
* Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
* Barrier methods of contraception: condom or occlusive cap. Use of oral, injected or implanted hormonal methods of contraception or other forms or hormonal contraception that have complete efficacy (failure less than 1 percent). (The dose of the contraceptive should be stable for 3 months)
* Active ongoing inflammatory diseases of the skin other than BP that might confound the evaluation of the benefit of Ixekizumab
* Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions) which, in the opinion of the investigator, significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy Investigator discretion should be used for subjects with pre-existing or recent-onset central or peripheral nervous system demyelinating disorders Significant medical problems, including but not limited to the following: uncontrolled hypertension, congestive heart failure (New York Heart Association (NYHA) status of class III or IV)
* Serum creatinine level exceeding 2.0 mg per dL (176.8 micro mol per L) at screening
* Total white blood cell (WBC) count less than 2,500 per microL, platelets less than 100,000 per microL, neutrophils less1500/microL or hemoglobin less than 8.5 g per dL, at screening
* Active systemic infections during the 2 weeks prior to randomization (common cold viruses not included) or any infection that reoccurs on a regular basis.
* Investigator discretion should be used regarding subjects who have traveled or resided in areas of endemic mycoses, such as histoplasmosis, coccidioidomycosis or blastomycosis and for subjects with underlying conditions that may predispose them to infection, such as advanced or inadequately controlled diabetes. Due to its endemic nature in Arizona, coccidioidomycosis screening is performed at baseline. A history of a disseminated coccidioidomycosis infection will exclude subjects.
* History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection as defined by a positive or indeterminate QuantiFERON Tuberculosis (TB)-Gold test (QFT) at screening.
* Subjects with a positive QFT test may participate in the study if a full tuberculosis work up (according to local practice/guidelines) is completed within 12 weeks prior to establishes conclusively that the subject has no evidence of active tuberculosis.

If the presence of latent tuberculosis is established, then treatment must have been initiated and maintained according to local country guidelines for at least 4 weeks prior to randomization.

* Past medical history of, or current infection with, human immunodeficiency virus (HIV), hepatitis B or hepatitis C prior to new diagnosis at screening
* History of lymphoproliferative disease and or any known malignancy and/or history of malignancy of any organ system within the past 5 years

Exceptions include:

For skin squamous cell carcinoma in situ and or well differentiate squamous cell carcinoma and/or basal cell carcinoma and or actinic keratosis and/or melanoma in situ that have been treated with no evidence of recurrence For the cervix carcinoma that has been removed For the colon non-invasive malignant colon polyps that have been removed

* Current severe progressive or uncontrolled disease which the investigator renders the subject unsuitable for the trial or puts the subject at increased risk Inability or unwillingness to undergo repeated venipuncture
* Any medical or psychiatric condition which, in the investigator's opinion, would keep the subject from adhering to the protocol or completing the study per protocol
* History or evidence of ongoing alcohol or drug abuse, within the last 6 months prior to the initiation of therapy
* Plans for administration of live vaccines during the study period or in the 12 weeks prior to the initiation of therapy
* Bacillus Calmette-Guerin (BCG) vaccination within 12 months of starting the study or with 12 months after completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Mangold, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixekizumab
Started | 4
Completed | 1
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ixekizumab
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (6.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Cessation of Blister Formation
Description: Median time to cessation of blister formation during the 12 weeks of therapy.
Time Frame: Up to 12 weeks
Population: Endpoint was not achieved as there was no cession of blisters.
Measure: Median (Standard Deviation); unit: days
Arm/Group | Ixekizumab
Number analyzed (Participants) | 4
days | NA (NA) — Insufficient number of participants with events.

2. Secondary Outcome: Change in Bullous Pemphigoid Disease Activity Index (BPDAI)
Description: The change in Bullous Pemphigoid Disease Activity Index (BPDAI) from week 0 to 12 of treatment will be measured.The BPDAI is a standard scoring system for cutaneous disease activity and pruritus in BP. BPDAI is predictive of the likelihood of a subsequent flare. The BPDAI consists of scoring various types of lesions and creates a score ranging from 0 to 120. A score of greater than 56 is considered severe disease.
Time Frame: Week 0 and week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ixekizumab
Number analyzed (Participants) | 4
units on a scale
  Week 0 | 24.8 (17.71)
  Week 12 | 39 (24.48)

3. Secondary Outcome: Prednisone Dose (mg)
Description: Average daily prednisone dose (mg) will be calculated for each Epoch.
Time Frame: Epoch 1 (washout- up to 4 weeks) Epoch 2 (week 0 to week 12) Epoch 3 (week 12 to week 16)
Population: Only one subject remained in the study by Epoch 3 timepoint (week 12 to 16)
Measure: Mean (Standard Deviation); unit: mg/d
Arm/Group | Ixekizumab
Number analyzed (Participants) | 4
mg/d
  Epoch 1 | 0 (0)
  Epoch 2 | 15.42 (9.17)
  Epoch 3: number analyzed (Participants) | 1
  Epoch 3 | 0 (0)

4. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0).
Description: The clinical safety of Ixekizumab will be monitored with collection of vital signs, clinical examination, and clinical laboratory studies. Adverse events (AE) will be reported per the Common Terminology Criteria for Adverse Events (CTCAEv4.0), a descriptive terminology which can be utilized for AE reporting. A grading (severity) scale is provided for each AE Grade refers to the severity of the AE. The CTCAE displays Grades 1-5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: weeks 0 to 18
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab
Number analyzed (Participants) | 4
Participants
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

5. Secondary Outcome: Decrease in Immunoglobulin G Anti-Bullous Pemphigoid 180 and 230 Antibody (Anti-BP180 & 230 IgG)
Description: We will measure the anti-BP180&230 antibodies through out treatment. These assays will be completed using and ELISA assay. Mayo medical labs references for anti-BP180&230 (<9.0 Units negative, > or = 9.0 Units positive)
Time Frame: week 0, 4, 8, 12
Population: This outcome measure was not achieved due to lack to sample to run assays.
Arm/Group | Ixekizumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Decrease in Neutrophil and Eosinophil Counts
Description: Neutrophil and eosinophil counts will be monitored throughout therapy. Mayo medical labs reports normal neutrophil levels (1.70-7.00X10(9)/L) and normal eosinophil levels (0.05-0.5X10(9)/L)
Time Frame: week 0, 4, 8, 12
Population: This outcome measure was not achieved due to lack of data.
Arm/Group | Ixekizumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Multiplex Cytokine Analysis
Description: Multiplex cytokine analysis will be performed throughout therapy on Interleukin (IL)- 6, 17, 22, 23, Transforming growth factor beta (TGFb), and matrix-metalloprotease-9 (MMP9).
Time Frame: week 0, 4, 8, 12
Population: This outcome measure was not achieved due to lack of sample to run assays.
Arm/Group | Ixekizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from baseline until 30 days post-study participation, for a total of approximately four to five months.
Arm/Group | Ixekizumab
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab (N=4)
Rib pain (General disorders) | 1 (1)
Skin Pain (General disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Staphylococcal overgrowth (Infections and infestations) | 1 (1)
Facial swelling (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT03099538/Prot_SAP_000.pdf